CLINICAL TRIAL: NCT04402125
Title: Reducing Stroke Risk in African-American Men
Acronym: TEAM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor, Case Western Reserve University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R01NR018023 (NIH); R01NR018023 (NIH)
Record Dates: First submitted 2020-05-15; First posted 2020-05-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Intervention Model Description: 80 participants are assigned to receive TEAM, and 80 participants are assigned to wait list
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants randomized to TEAM intervention for 6 months, then observed for 6 month follow up
  Interventions: Behavioral: TargEted MAnageMent Intervention (TEAM)
- Waitlist (Other): Participants randomized to waitlist for 6 months, then offered the intervention for 6 months
  Interventions: Behavioral: TargEted MAnageMent Intervention (TEAM)

INTERVENTIONS:
Behavioral: TargEted MAnageMent Intervention (TEAM) — TEAM targets acquisition of self-management expertise and use of healthy behaviors that are intended to reduce stroke risk and burden. TEAM participants will continue in their regular medical care, supplemented by the TEAM intervention. Components are as follows:
  1. A 60 minute initial session in which the nurse and the PED meet with the patient who has experienced stroke or TIA. The initial session will cover introductions, orientation, and logistic planning.
  2. Five 60-minute group sessions with 6-10 stroke survivors (and their care partners as applicable) held approximately 4 weeks, 6 weeks, 8 weeks, 10 weeks, and 12 week after enrollment. Sessions are co-lead by a nurse and a PED.
  3. Six brief telephone sessions implemented after the conclusion of the 5 TEAM group sessions. Calls will be conducted every 2 weeks for 12 weeks. Calls will reinforce group session content, provide social support and facilitate linkage with other care providers.

SUMMARY:
The project is a 6-month prospective Randomized Controlled Trial evaluating the effects of TargEted MAnageMent Intervention (TEAM, N=80) vs. wait-list (WL, N=80) control in African American men who have experienced a stroke or TIA within the past 5 years.

DETAILED DESCRIPTION:
The project is a 6-month prospective Randomized Controlled Trial evaluating the effects of TargEted MAnageMent Intervention (TEAM, N=80) vs. wait-list (WL, N=80) control in African American men who have experienced a stroke or TIA within the past 5 years. TEAM features a nurse-led, person-centered, holistic intervention that takes advantage of existing strengths in AA families/communities. TEAM uses peer educator dyads (PEDs) to provide support and model behaviors. The PED consists of an AA man peer educator (PE) with experience in managing his own stroke risk and a care partner. A care partner is someone who is the family member, friend or other individual of someone who has had a stroke or TIA. A care partner can be associated with a PE but they do not have to be. PEs and care partners will be matched depending on schedules and availability and may not always be members of the same household. The nurse and PED co-deliver TEAM to an AA male patient who has experienced stroke or TIA. Patients are also encouraged to include a family, friend, or other individual important his stroke recovery in the TEAM programming. The intervention is a practical approach suitable for implementation in specialty, primary care or community settings, and has the potential to reverse the unacceptably high morbidity seen in AA men due to stroke-related disorders.

ELIGIBILITY:
Inclusion Criteria for RCT participant:

1. Age range 18 to 90
2. Self-identified African American male
3. Have had a stroke or TIA in the past 10 years based on date of hospital discharge from an acute stroke program or Emergency Room/physician visit for TIA
4. Barthel Index (BI) score of >= 40
5. Able to participate in group sessions

Inclusion Criteria for Care Partner

1. Age range from 18 to 90
2. Able to participate in group sessions

Inclusion criteria for peer educator:

1. Age range: from 18 to 90
2. Self-identified African American male
3. Have had a stroke or TIA
4. Able to participate in group sessions

Inclusion Criteria for Peer Educator Care Partner

1. Age range: from 18 to 90
2. Able to participate in group sessions
3. Is either a family member, friend or other individual who is important in an enrolled peer educator's stroke recovery OR the family member, friend or other individual of someone who has had a stroke or TIA and is/was important in their stroke recovery

Exclusion Criteria for RCT participant

1. Individuals who are unable or unwilling to provide written informed consent
2. Individuals who have had stroke due to sickle-cell disease

Exclusion Criteria for Care Partner participant 1. Individuals who are unable or unwilling to provide written informed consent

Exclusion Criteria for Peer Educator

1. Individuals who are unable or unwilling to provide written informed consent
2. Individuals who have had stroke due to sickle-cell disease

Exclusion Criteria for Peer Educator's Care Partner

1. Individuals who are unable or unwilling to provide written informed consent

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
TEAM vs WL change in systolic BP | Baseline to 6-month follow up
  TEAM vs WL change in systolic BP

SECONDARY OUTCOMES:
TEAM vs WL change in diastolic BP | Baseline to 6-month follow up
  TEAM vs WL change in diastolic BP
TEAM vs WL change in cholesterol | Baseline to 6-month follow up
  TEAM vs WL change in cholesterol
TEAM vs WL change in HDL | Baseline to 6-month follow up
  TEAM vs WL change in HDL
TEAM vs WL change in LDL | Baseline to 6-month follow up
  TEAM vs WL change in LDL
TEAM vs WL change in triglycerides | Baseline to 6-month follow up
  TEAM vs WL change in triglycerides
TEAM vs WL change in BMI | Baseline to 6-month follow up
  TEAM vs WL change in BMI
TEAM vs WL change in HbA1c | Baseline to 6-month follow up
  TEAM vs WL change in HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Still CH, Burant C, Moore S, Einstadter D, Killion C, Modlin C, Sundararajan S, Thornton JD, Wright JT Jr, Sajatovic M. The Targeted Management (TEAM) Intervention for Reducing Stroke Risk in African American Men: Rationale and Study Design of a Prospective Randomized Controlled Trial. J Multidiscip Healthc. 2021 Feb 23;14:513-522. doi: 10.2147/JMDH.S288753. eCollection 2021. PMID 33654407